CLINICAL TRIAL: NCT02304185
Title: A First in Human Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Dose Levels of Trimeric gp140 Protein in Healthy Adult Volunteers
Brief Title: Safety, Tolerability and Immunogenicity Study of 2 Dose Levels of Trimeric Glycoprotein140 (gp140) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR104488; HIV-V-A003 (Other: Crucell Holland BV); IPCAVD008 (Other: Crucell Holland BV)
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Healthy; Acquired Immuno-Deficiency Syndrome; Acquired Immunodeficiency Syndrome Virus; Glycoprotein; Adjuvant; Vaccine; Placebo
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — GP 140; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- gp140, 50 mcg (Experimental)
  Interventions: Biological: gp140, 50 mcg
- gp140, 50 mcg + Adjuvant (Experimental)
  Interventions: Biological: gp140, 50 mcg + Adjuvant
- Placebo 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- gp140, 250 mcg (Experimental)
  Interventions: Biological: gp140, 250 mcg
- gp140, 250 mcg + Adjuvant (Experimental)
  Interventions: Biological: gp140, 250 mcg + Adjuvant
- Placebo 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: gp140, 50 mcg — Glycoprotein 140 (gp140) vaccine containing 50 microgram (mcg) total protein will be administered intramuscularly on Day 1 and Day 29.
  Arms: gp140, 50 mcg
Biological: gp140, 50 mcg + Adjuvant — The gp140 vaccine containing 50 mcg total protein mixed with 0.425 milligram (mg) aluminum phosphate adjuvant will be administered intramuscularly on Day 1 and Day 29.
  Arms: gp140, 50 mcg + Adjuvant
Biological: gp140, 250 mcg — The gp140 vaccine containing 250 mcg total protein will be administered intramuscularly on Day 1 and Day 29.
  Arms: gp140, 250 mcg
Biological: gp140, 250 mcg + Adjuvant — The gp140 vaccine containing 250 mcg total protein mixed with 0.425 mg aluminum phosphate adjuvant will be administered intramuscularly on Day 1 and Day 29.
  Arms: gp140, 250 mcg + Adjuvant
Drug: Placebo — Placebo matched to gp 140 vaccine drug product will be administered intramuscularly on Day 1 and Day 29.
  Arms: Placebo 1; Placebo 2

SUMMARY:
The purpose of this study is to assess the safety and tolerability of 2 different dose levels of trimeric glycoprotein140 (gp140) administered as a 2-dosage regimen, intramuscularly (injection of a substance into a muscle), with and without aluminum phosphate as adjuvant in healthy human immunodeficiency virus (HIV)-uninfected participants.

DETAILED DESCRIPTION:
This is a single-center, randomized (the study drug is assigned by chance), placebo-controlled (study in which the experimental treatment or procedure is compared to a pretend treatment with no drug in it to test if the drug has a real effect), and double-blind (neither physician nor participant knows the treatment that the participant receives) study. The study comprises a Screening Period (up to 4 weeks), a Vaccination Period (participants will be vaccinated on Days 1 and 29), and a Follow-up Period (up to 48 weeks). All eligible participants will be randomly assigned to 1 of the 2 sequential cohorts (low dose cohort and high dose cohort). Participants in low dose cohort will receive 1 of the following treatments: low dose (50 microgram [mcg]) gp140 drug product (DP), low dose gp140 DP with adjuvant (aluminum phosphate), placebo matched to low dose DP; and participants in high dose cohort will receive 1 of the following treatments: high dose (250 mcg) gp140 DP, high dose gp140 DP with adjuvant, and placebo matched to high dose DP. There will be an interim safety review of safety/tolerability from low-dose cohort before the high-dose cohort receives study treatment. Total study duration will be 56 weeks per participant. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical examination, medical history, electrocardiogram (ECG), laboratory criteria, and vital signs measurement performed at Screening
* Participants are negative for human immunodeficiency virus (HIV) infection at Screening (negative United States Food and Drug Administration-approved HIV diagnostic blood test)
* All female participants of childbearing potential must have a negative serum (beta human chorionic gonadotropin) at Screening, and a negative urine pregnancy test pre-dose on Day 1 and Day 29
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction until 3 months after receiving the last dose of study vaccine. A man must agree not to donate sperm until 3 months after receiving the last dose of study vaccine
* Participants are assessed by the clinic staff as being at low risk for HIV infection

Exclusion Criteria:

* Participant has chronic active hepatitis B or active hepatitis C, active syphilis infection, chlamydia, gonorrhea, or trichomonas. Active syphilis documented by exam or serology unless positive serology is due to past treated infection
* In the 12 months prior to enrollment, participant has a history of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranulomavenereum, chancroid, or hepatitis B
* Participant has any clinically significant acute or chronic medical condition that in the opinion of the Investigator would preclude participation (for example, history of seizure disorders, bleeding/clotting disorder, autoimmune disease, active malignancy, poorly controlled asthma, active tuberculosis or other systemic infections)
* Participant has had major surgery within the 4 weeks prior to study entry or planned major surgery through the course of the study
* Participant has had a thyroidectomy, or thyroid disease requiring medication during the last 12 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Local and Systemic Reactogenicity Events Over 8 Days After First Vaccination | Day 8
  Participants will be asked to note occurrences of local reactions: erythema, induration, swelling, pain/tenderness, itching, or warmth at the injection site, and systemic events: daily temperature, fatigue, headache, myalgia, arthralgia, chills, nausea, vomiting, rashes, and general itching daily for 8 days post-vaccination. These occurrences will be recorded through the memory aid provided to serve as a reminder to the participants for the next clinic visit.
Number of Participants With Local and Systemic Reactogenicity Events Over 8 Days After Second Vaccination | Day 36
  Participants will be asked to note occurrences of local reactions: erythema, induration, swelling, pain/tenderness, itching, or warmth at the injection site, and systemic events: daily temperature, fatigue, headache, myalgia, arthralgia, chills, nausea, vomiting, rashes, and general itching daily for 8 days post-vaccination. These occurrences will be recorded through the memory aid provided to serve as a reminder to the participants for the next clinic visit.
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Week 52 or early withdrawal
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Envelop (Env) Binding Antibody Titer at Week 8 | Week 8
  The humoral immune response will be assessed by Env Clade C-specific enzyme-linked immunosorbent assay (ELISA) binding antibody titer at Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trials, Study Director — Crucell Holland BV
Locations (1):
- Miami, Florida, United States